CLINICAL TRIAL: NCT00174616
Title: Phase 2 Study of Weekly Oxaliplatin and Capecitabine (XELOX) in Combination With Preoperative Radiotherapy in Patients With MRI Defined Locally Advanced Rectal Cancer
Brief Title: CORE: Capecitabine, Oxaliplatin, Radiotherapy and Excision
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C_8601
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Oxaliplatin, capecitabine, radiotherapy

INTERVENTIONS:
Drug: Oxaliplatin, capecitabine, radiotherapy — * Oxaliplatin 50mg/m² I.V. 2 hours weekly x 5 doses
  * Capecitabine 825mg/m² P.O. B.I.D. daily x 5 days x 5 weeks
  * Radiotherapy 45 Gy total (1.8Gy/dose) 25 fractions daily x 5 days x 5 weeks

SUMMARY:
Primary objective:

* Pathological complete response (ypT0N0) rate

Secondary objectives:

* Histopathological R0 resection rate
* Pathological downstaging (ypT0-T2N0) rate
* One month surgical complication rate
* Predictive value of pre-operative MRI for surgical, pathological and clinical outcomes
* Safety
* Local and distant recurrence rates
* Progression-free survival
* Overall survival

ELIGIBILITY:
* Histologically proven adenocarcinoma of the rectum (Tumour ≤ 12 cm from the anal verge)
* No evidence of distant spread
* No prior therapy for chemotherapy or radiation therapy for rectal cancer
* Patient considered locally advanced by MRI:

  * Tumour beyond mesorectal fascia, or
  * Tumour ≤ 2mm from mesorectal fascia, or
  * T3 tumour < 5cm from anal verge
* For female patient of childbearing potential, neither pregnant nor breastfeeding, and under active contraception
* No peripheral neuropathy > grade1
* ECOG PS ≤ 2
* ANC > 1,500 x 10^9/L
* Platelets > 100,000 x 10^9/L
* Creatinine < 1.5 x IULN
* Bilirubin < 1.5 IULN
* SGPT (ALT) < 2.5 IULN
* No pre-existing condition which would deter chemoradiotherapy
* No uncontrolled diarrhoea or fecal incontinence
* No significant small bowel (> 200cc or 6X6X6cm) delineated within the radiation fields
* No other serious uncontrolled concomitant illness
* Informed consent signed

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2003-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
MRI staging and TME surgery | within 4 - 6 weeks after completion XELOX-RT

SECONDARY OUTCOMES:
Measure safety - NCI-CTC version 2 | from baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Pe Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom